CLINICAL TRIAL: NCT06283667
Title: A Multi-centre, Prospective, Non-interventional, Single-armed, 104 Weeks Post-marketing Study to Investigate Safety and Clinical Parameters of Wegovy® Once Weekly in Patients With Obesity Disease Under Real-world Clinical Practice Conditions
Brief Title: Special Use - Results Surveillance on Long-term Use With Wegovy®
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-4872; U1111-1266-3863 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wegovy®: Patients with obesity treated with Wegovy® (semaglutide) once weekly under real-world clinical practice conditions in Japan.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Paricipants will be treated with commercially available Wegovy® according to routine clinical practice at the discretion of the treating physician, following approved label in Japan. The decision to initiate treatment with commercially available Wegovy® has been made by the patient and the treating physician before and independently from the decision to participate in this study.
  Other Names: Wegovy®

SUMMARY:
The purpose of the study is to investigate the safety and effectiveness of Wegovy® in patients with obesity disease under real-world clinical practice in Japan. Participants will get Wegovy® as prescribed by the study doctor. The study will last for about 4 years. Participant will be in the study for about 2 years (104 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* The decision to initiate treatment with commercially available Wegovy® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study
* Male or female, no age limitation
* Diagnosis of obesity disease; with either hypertension, dyslipidaemia or type 2 diabetes, insufficiently controlled with diet and exercise therapies, and should meet either of:

  1. Body mass index (BMI)* greater than or equal to 27 kilograms per meter square (kg/m^2) with two or more obesity-related comorbidities**, or
  2. BMI* greater than or equal to 35 kg/m^2
* Participant who has never been exposed to Semaglutide or who started treatment with Wegovy® within the past 4 weeks at registration

  * BMI calculation will be based on height and body weight recorded in the enrolment form of electronic case report form (eCRF) at enrolment.

    * Definition of obesity-related comorbidities are in accordance with Japan Student Services Organization (JASSO) guideline 3: (1) impaired glucose tolerance, (2) dyslipidaemia, (3) hypertension, (4) hyper-uricemia/gout, (5) coronary artery disease, (6) cerebral infarction, (7) non-alcoholic fatty liver disease, (8) menstrual disorder/infertility, (9) obstructive sleep apnoea syndrome/obesity-hypoventilation syndrome, (10) locomotory disease or (11) obesity-related kidney disease.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Treatment with any investigational drug within 30 days prior to baseline (Visit 1)
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* A history of hypersensitivity to any ingredients of this drug
* Diabetic ketoacidosis, diabetic coma, pre-coma or type 1 diabetes mellitus [The treatment with insulin is mandatory. It is not appropriate to use this drug]
* In emergency cases such as severe infections and surgery in patients with type 2 diabetes [It is desirable to control blood glucose with insulin; therefore, administration of this drug is not appropriate]
* Pregnant or possibly pregnant female
* Female who plans to become pregnant within 2 months

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants are patients with obesity treated with Wegovy® (semaglutide) once weekly under real-world clinical practice conditions in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Reactions (ARs) | From baseline (week 0) to end of study (week 104)
  Measured as count of events

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | From baseline (week 0) to end of study (week 104)
  Measured as count of events
Number of serious adverse events (SAEs) | From baseline (week 0) to end of study (week 104)
  Measured as count of events
Number of Serious Adverse Reactions (SARs) | From baseline (week 0) to end of study (week 104)
  Measured as count of events
Change in body weight (Percent (%)) | From baseline (week 0) to end of study (week 104)
  Measured as percent (%)
Change in body weight (Kilograms (Kg)) | From baseline (week 0) to end of study (week 104)
  Measured in kilograms (Kg)
Change in waist circumference | From baseline (week 0) to end of study (week 104)
  Measured in centimeters (cm)
Change in BMI (Body Mass Index) | From baseline (week 0) to end of study (week 104)
  Measured in kilogram per meter square (kg/m^2)
Change in body weight after treatment discontinuation | From treatment discontinuation after at least 12 weeks to end of study (week 104)
  Measured as percent (%)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (112):
- Japan (111):
  - Novo Nordisk Investigational Site, Tokyo, Chiyoda City
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Okazaki City Hospital, Aichi
  - Nagoya City University Hospital_Obesity Treatment Center, Aichi
  - Fujita Health University Hospital_Endocrinology, Diabetes and Metabolism, Aichi
  - Ichinomiyanishi Hospital, Aichi
  - Nakadori General Hospital_Diabetes and Endocrinology, Akita
  - Odate Municipal General Hospital_Endocrinology and Metabolism, Akita
  - Akita University Hospital, Diabetes and Endocrinology, Akita-shi, Akita
  - Hachinohe City Hospital_Diabetes and Metabolism, Aomori
  - Juntendo University Hospital_Tokyo, Bunkyo-ku, Tokyo
  - Shinmatsudo Central General Hospital_Diabetes and Endocrinology, Chiba
  - Toho University Medical Center Sakura Hospital, Chiba
  - Kimitsu Chuo Hospital_Diabetology and Endocrinology, Chiba
  - Kameda Medical Center_Diabetes and Endocrinology, Chiba
  - Fukuoka University Chikushi Hospital_Endocrinology and Diabetes Mellitus, Chikushino-shi, Fukuoka
  - Chiba University Hospital_Diabetes, Metabolism and Endocrinology, Chiyoda-ku, Tokyo
  - Mikannohana Clinic, Ehime
  - Matsuyama Shimin Hospital_Diabetes and Endocrinology, Ehime
  - University of Fukui Hospital, Fukui
  - National Hospital Organization Fukuokahigashi Medical Center, Fukuoka
  - Fukuoka Kieikai Hospital_Diabetes and obesity centre, Fukuoka
  - Fukuoka Sanno Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka-shi, Fukuoka
  - Fukushima Medical University Hospital_Diabetes and Endocrinology, Fukushima
  - Chuno Kosei Hospital_Endocrinology and Diabetes, Gifu
  - Matsunami General Hospital_Diabetes and Endocrinology, Gifu
  - Ogaki Municipal Hospital_Diabetes and Nephrology, Gifu
  - Gunma University Hospital, Dept. of Endocrinology and Diabetes, Gunma
  - Hamamatsu University Hospital, Hamamatsu-shi, Shizuoka
  - Murakami Memorial Hospital_Diabetes Internal Medicine, Hiroshima
  - Mazda Hospital_Diabetes, Hiroshima
  - Sapporo Tonyobyo Kojosen Clinic, Hokkaido
  - Japanese Red Cross Asahikawa Hospital, Hokkaido
  - Hyogo Medical University Hospital_Diabetes, Endocrinology and Metabolism, Hyōgo
  - University of Tsukuba Hospital_Diabetes and Endocrinology, Ibaraki
  - Shimane Univ. HP, Dept of Endocrinology&Metabolism, Izumo, Shimane
  - Kagoshima University Hospital_Diabetes and Endocrinology, Kagoshima
  - Kawasaki Municipal Hospital_Diabetes and Endocrinology, Kanagawa
  - Kanto Rousai Hospital_Diabetes and Endocrinology, Kanagawa
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Yokohama Rosai Hospital_Diabetes and Endocrinology, Kanagawa
  - Showa University Fujigaoka Hospital_Internal Medicine, Kanagawa
  - Yokohama City Minato Red Cross Hospital_Endocrinology, Kanagawa
  - Yokohama City University Medical Center_Endocrinology and Diabetes, Kanagawa
  - Tokai University Hospital_Nephrology, Endocrinology and Metabolism, Kanagawa
  - Yokohama City University Medical Center_Nephrology and Hypertension, Kanahawa
  - Kasugai Municipal Hospital_Cardiovascular Medicine, Kasugai-shi, Aichi
  - Nippon Medical School Musashikosugi Hospital_Neurological Surgery, Kawasaki-shi, Kanagawa-ken
  - Kochi Medical School Hospital_Endocrinology, Metabolism and Nephrology, Kochi
  - Kumamoto General Hospital_Diabetes Center, Kumamoto
  - Minamata City General Hospital & Medical Center_Metabolism, Kumamoto
  - Kumamoto University Hospital, Diabetes, Metabo and Endo, Kumamoto-shi, Kumamoto
  - Kure Medical Center and Chugoku Cancer Center, Kure-shi, Hiroshima
  - Shin Koga Hospital, Kurume-shi, Fukuoka
  - University Hospital Kyoto Prefectual University of Medicine, Kyoto
  - Kyoto City Hospital_Diabetes and Metabolism, Kyoto
  - Kyoto University Hospital, Kyoto-shi, Kyoto
  - National Hospital Organization Kyoto Medical Center_Cardiology, Kyoto-shi, Kyoto
  - Mie University Hospital_Mie, Mie
  - Japanese Red Cross Ise Hospital_Diabetes and Metabolism, Mie
  - Miura Central Clinic, Miura-shi, Kanagawa
  - Aichi Medical University Hospital, Diabetes Medicine, Nagakute-shi, Aichi
  - Nagano Matsushiro General Hospital_department of diet, Nagano
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa-ken
  - Iwate Medical University Uchimaru Medical Center, Division of Diabetes and Metabolism and Endocrine medicine, Numakunai
  - Okayama University Hospital_Neph. and Diabetes, Metabolism, Okayama
  - Okayama Rosai Hospital_Cardiology, Okayama
  - Okayama Medical Center_Cardiology, Okayama-shi, Okayama
  - Urasoe General Hospital_Cardiology, Okinawa
  - Osaka National Hospital_Osaka, Osaka
  - Osaka Metropolitan University Hospital_Lifestyle disease diabetes centre, Osaka
  - Chibune Hospital_Diabetes and Endocrinology, Osaka
  - Matsushita Memorial Hospital_Diabetes and Endocrinology, Osaka
  - Kishiwada City Hospital_Endocrinology and Metabolism, Osaka
  - Bellland Sogo Byoin_Endocrinology and Metabolism, Osaka
  - Osaka City General Hospital_Endocrinology and Diabetes Mellitus, Osaka-shi, Osaka
  - Osaki citizen hospital_Diabetes and metabolic disease, Osaki-shi, Miyagi
  - Shinbeppu Hospital_Endocrinology and Metabolism, Ōita
  - Karatsu Redcross Hospital_Diabetes Internal Medicine, Saga
  - NTT East Japan Sapporo HP_Diabetes Mellitus & Int med Endo, Sapporo, Hokkaido
  - Sapporo Medical University Hospital_Cardiovascular, Kidney, Metabolism Endocrinology, Sapporo-shi, Hokkaido
  - Aso Clinic, Shizuoka
  - Juntendo University Shizuoka Hospital_Diabetes and Endocrinology, Shizuoka
  - JA Shizuoka Kohseiren Enshu Hospital_Internal Medicine, Shizuoka
  - Hamamatsu Medical Center, Shizuoka
  - Japanese Red Cross Hamamatsu Hospital_Cardiology, Shizuoka
  - Chutoen General Medical Center_Diabetes and Endocrinology, Shizuoka
  - Nagasaki Hospital_Internal Medicine, Tochigi
  - Sano Kosei General Hospital_Neph.& Endocrinology,Metab., Tochigi
  - Tamaki Aozora Byoin_Diabetes and Endocrinology, Tokushima
  - Gifu University Hospital, Tokyo
  - Nihon University Hospital_Internal Medicine, Tokyo
  - Tokyo Teishin Hospital, Tokyo
  - Nihonbashi Leiwa Naika Clinic, Tokyo
  - The Jikei University Hospital Dept of Diabetes, Metabolic, Tokyo
  - Institute of Science Tokyo Hospital_Cardiology, Tokyo
  - National Center for Child Health and Development_Internal medicine for women, Tokyo
  - Keio University Hospital, Tokyo
  - Tokyo Women's Medical University_Diabetes and Metabolism, Tokyo
  - Kyorin University Hospital_Diabetes and Endocrinology, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Tokyo
  - Tottori University Hospital_Endocrinology and Metabolism, Tottori
  - Tottori University Hospital_Pharmacotherapy, Tottori
  - Toyohashi Municipal Hospital, Toyohashi-shi, Aichi-ken
  - Japanese Red Cross Wakayama Medical Center_Diabetology and Endocrinology, Wakayama
  - Wakayama Medical Univercity Hospital_Diabetes and Endocrinology, Wakayama
  - Yamagata University Hospital, Internal Medicine 3, Yamagata-shi, Yamagata
  - Shimonoseki Medical Center_Diabetes and Endocrinology, Yamaguchi
  - Yamaguchi Rosai Hospital_Diabetes and Endocrinology, Yamaguchi
  - Yokohama City University Hospital, Endocrinology, Metabolism, Yokohama, Kanagawa
- Tokyo Medical Univ. Hospital_Diabetes, Metabolism and Endocrinology

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com